CLINICAL TRIAL: NCT00155272
Title: A Pilot Clinical and Mechanistic Study of Radiotherapy Plus Thalidomide in Locally Advanced Hepatocellular Carcinoma
Brief Title: Radiotherapy Plus Thalidomide in Locally Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 931003
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Radiotherapy; Thalidomide; Dynamic contrast enhanced MRI
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
This is a pilot study of concomitant radiotherapy and thalidomide for patients with locally advanced HCC.Besides toxicity and efficacy, mechanistic studies including dynamic contrast enhanced MRI and serum cytokines will be evaluated.

DETAILED DESCRIPTION:
This is a pilot study of concomitant radiotherapy and thalidomide for patients with locally advanced HCC. Patients whose tumor(s) are not suitable for other local treatment, such as surgery, trans-arterial chemoembolization (TAE), ethanol injection, or radiofrequency ablation. will be enrolled.Radical radiotherapy will be started after pre-treatment evaluation. The total dose of RT will be 50Gy in 25 fractions to local tumor(s). Oral Thalidomide will be started 3 days before RT begins. Thalidomide treatment will continue for totally 6 months or until tumor progression. Dynamic contrast enhanced MRI (DCEMRI) will be done at the following time points to assess the change in tumor perfusion: (1) before the start of thalidomide treatment; (2) 3 days after thalidomide before radiotherapy; (3) 2weeks after radiotherapy begins;and (4) 1 month after radiotherapy completes. DCEMRI will then be done every 3 months until disease progression.Serum samples for angiogenic cytokine studies will also be collected.The study was designed to evaluate the feasibility and tolerability of combination treatment of radiotherapy and thalidomide for locally advanced HCC. The sample size was determined by the expected incidence of grade 4 toxicity of the combination treatment versus radiotherapy alone for locally advanced HCC. Since the grade 4 toxicity of radiotherapy alone is 7-9%, we need at least 15 patients to evaluate for feasibility of the combination treatment. With an estimated drop out rate of approximately 10%, 17 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1.1 Patients with measurable, locally advanced HCC that are not suitable for other local therapies, including surgery, TAE, alcohol injection, or radiofrequency ablation.

1.2 Patients with histological confirmed HCC or patients who do not have histological diagnosis but have met all of the following criteria: 1.2.1 Presence of chronic viral hepatitis and/or cirrhosis 1.2.2 Presence of hepatic tumor(s) with image findings (sonography, CT scan) compatible with HCC.

1.2.3 A persistent elevation of serum a-fetoprotein level ³ 400 ng/ml without any evidence of ana-fetoprotein-secreting germ cell tumor.

1.3 Patients without any local or systemic therapy for HCC within 4 weeks. 1.4 Patients with age > 20 years and < 70 years. 1.5 Patients with a performance status of ECOG score < 1. 1.6 Patients must fulfill all of the following criteria: 1.6.1 Child-Pugh's Score ≦ 7. 1.6.2 Serum total bilirubin < 1.5 times upper normal limit (UNL 1.6.3 Serum alanine transaminase (ALT) < 5 times UNL 1.6.4 Platelet count > 5.0 x 104 / mm3. 1.6.5 White blood cell count > 3,000 / mm3. 1.6.6 Serum creatinine < 2.0 mg/dL 1.7 Patient must have local tumors less than one half of the whole liver and the tumors can be encompassed within RT fields 1.8 Signed informed consent 1.9 Sexually active patients, in conjunction with their partner, must practice birth control during, and for 2 months after, thalidomide therapy.

1.10 Female patients in child-bearing age must have negative pregnancy test.

Exclusion Criteria:

* 2.1. Patients with documented extrahepatic metastasis. 2.2. Patients who received previous radiotherapy to abdominal area. 2.3. Patients who have received thalidomide treatment prior to enrollment. 2.4. Patients who had other investigational drug treatment within 4 weeks prior to enrollment.

2.5. Patients with NCI grade 2 or greater peripheral neuropathy of any causes. 2.6. Patients with other systemic diseases that required concurrent usage of glucocorticosteroid or immunosuppressant agent(s).

2.7. Patients who have major systemic diseases that the attending physicians consider inappropriate for radiotherapy or thalidomide therapy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19
Dates: Start 2005-03; Study Completion 2005-08

PRIMARY OUTCOMES:
The primary endpoint is the feasibility and tolerability of thalidomide plus radiotherapy.

SECONDARY OUTCOMES:
The secondary end point is correlation of parameters of tumor perfusion assessed by DCEMRI and serum cytokine levels with objective tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ju Ch'ang, M.D., Principal Investigator — National Health Research Institutes, Division of Cancer Research; Chih-Hung Hsu, M.D., Study Chair — National Taiwan University Hospital; Tiffany Ting Fang Shih, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan

REFERENCES:
- [Derived] Liang PC, Ch'ang HJ, Hsu C, Chen LT, Shih TT, Liu TW. Perfusion parameters of dynamic contrast-enhanced magnetic resonance imaging predict outcomes of hepatocellular carcinoma receiving radiotherapy with or without thalidomide. Hepatol Int. 2015 Apr;9(2):258-68. doi: 10.1007/s12072-014-9557-1. Epub 2014 Jul 26. PMID 25788178
- [Derived] Ch'ang HJ, Hsu C, Chen CH, Chang YH, Chang JS, Chen LT. Phase II study of concomitant thalidomide during radiotherapy for hepatocellular carcinoma. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):817-25. doi: 10.1016/j.ijrobp.2010.10.067. Epub 2011 Jan 27. PMID 21277098